CLINICAL TRIAL: NCT02757508
Title: Healthy and Affordable Protein Rich Foods for African Market School Feeding Programs
Brief Title: Healthy and Affordable Protein Rich Foods for African Market
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: University of Ghana (Other); Arla Foods (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Other
Other Study IDs: HAPFAM
Record Dates: First submitted 2016-04-20; First posted 2016-05-02 (Estimated); Last update posted 2018-02-13 (Actual); Status verified 2018-02

CONDITIONS: School Feeding Programs and Nutrition Supplements
MeSH Terms: interventions — Vitamins; Minerals

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Control (Active Comparator): Vitamins/minerals-200 mg premix
  Interventions: Dietary Supplement: Vitamins/minerals
- Group 1 (Experimental): Vitamins/minerals + Milk Protein (8.75 g)-the milk protein is a skim milk powder with the sugar lactose.
  Interventions: Dietary Supplement: protein powder supplement
- Group 2 (Experimental): Vitamins/minerals + Milk/plant Protein (8.75g)-the milk protein is a skim milk protein powder and the plant protein is a rice protein concentrate and the sugar lactose.
  Interventions: Dietary Supplement: protein powder supplement
- Group 3 (Experimental): Vitamins/minerals + Milk Protein (4.38g)-the milk protein is a skim milk protein powder with the sugar lactose.
  Interventions: Dietary Supplement: protein powder supplement

INTERVENTIONS:
Dietary Supplement: protein powder supplement
  Arms: Group 1; Group 2; Group 3
Dietary Supplement: Vitamins/minerals
  Arms: Control

SUMMARY:
This study is to gather information on school feeding programs and to measure the effect on linear growth and cognitive performance when providing a high-quality milk protein source or a combination of a high-quality milk protein source and rice proteins as a nutritional supplement to school children in Ghana. Children will receive a meal with a protein powder supplement with vitamins and minerals mixed into it. Participation is expected to last for 9 months.

1200 Children aged 6-7 years attending school will be enrolled throughout twenty primary schools (60 per school). Participants will be randomized to one of four groups: Control: Vitamins/minerals-200 mg premix contain the required micronutrients as per UNICEF recommendations.

For groups 1-3 the same vitamin/mineral mix will be used along with Group 1. Vitamins/minerals + Milk Protein (8.75 g)-the milk protein is a skim milk powder with the sugar lactose.

Group 2. Vitamins/minerals + Milk/plant Protein (8.75g)-the milk protein is a skim milk protein powder and the plant protein is a rice protein concentrate and the sugar lactose.

Group 3. Vitamins/minerals + Milk Protein (4.38g)-the milk protein is a skim milk protein powder with the sugar lactose.

At baseline measurements-weight,height,mid-upper arm circumference,and body composition will be taken, fasting blood spot test will be administered to measure levels of Insulin and insulin like growth factor and other metabolic test, and computer based cognitive testing. Demographic information will be collected along with a dietary survey. Primary outcomes are cognitive performance on standardized tests and change in height-for-age z-score over the supplementation period, 9 months total. Questionnaires will be administered to collect demographic data and dietary information.

At the mid-point all measurements will be taken again and cognitive testing will be repeated.

At the end of the study all measurements will be taken again, cognitive testing repeated, blood spot samples taken again, and a short survey will be administered about the protein powders.

ELIGIBILITY:
Inclusion Criteria:

* Ghana school children between the ages of 6-9 years old

Exclusion Criteria:

* children with severe malnutrition
* chronic debilitation disease
* milk allergy

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1041 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2017-07-30 (Actual); Study Completion 2017-07-30 (Actual)

PRIMARY OUTCOMES:
Cognitive performance on Cambridge Cognition tests (CANTAB) | 9 months
  Five tests created by Cambridge Cognition (CANTAB) will be selected and administered at enrollment, halfway through the intervention, and at the end of the intervention. The tests will examine visual memory pattern, recognition memory, test comprehension, rule acquisition, and attention set shifting. These tests will be administered on a Windows tablet by trained research staff. The participants will start by taking a practice test to get use to using the tablet and test format.
Change in height-for-age z score over the period of supplementation. | 9 months

CONTACTS AND LOCATIONS:
Locations (2):
- Washington University School of Medicine, St Louis, Missouri, United States
- Atebubu, Ghana

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual data available

REFERENCES:
- [Derived] Lee R, Singh L, van Liefde D, Callaghan-Gillespie M, Steiner-Asiedu M, Saalia K, Edwards C, Serena A, Hershey T, Manary MJ. Milk Powder Added to a School Meal Increases Cognitive Test Scores in Ghanaian Children. J Nutr. 2018 Jul 1;148(7):1177-1184. doi: 10.1093/jn/nxy083. PMID 29905824